CLINICAL TRIAL: NCT06870591
Title: Pivotal Method-Comparison Study for the Cardiac Performance System (CPS) to Measure Hemodynamic Parameters
Brief Title: Pivotal Study for the Cardiac Performance System (CPS)
Status: Recruiting | Type: Observational
Sponsor: Sensydia Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CPS_PIVOTAL
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac Performance System; CPS; Hemodynamic Parameters; Right Heart Catheterization
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CPS Measurement Group: Participants undergoing clinically indicated right heart catheterization will receive a single, non-invasive measurement using the Cardiac Performance System (CPS) before their scheduled procedure. The study aims to compare CPS results with standard invasive hemodynamic measurements.
  Interventions: Device: Cardiac Performance System (CPS)

INTERVENTIONS:
Device: Cardiac Performance System (CPS) — CPS is a non-invasive platform for hemodynamic assessment that uses acoustic sensors and electrocardiogram electrodes.

SUMMARY:
This multi-center, observational study evaluates the accuracy of the Cardiac Performance System (CPS), a non-invasive device, for measuring hemodynamic parameters in adult patients undergoing clinically indicated right heart catheterization. The study compares CPS measurements to invasive measurements to assess agreement and potential clinical utility.

DETAILED DESCRIPTION:
The study will enroll adults undergoing right heart catheterization as part of their clinical care. A single CPS measurement will be performed before the scheduled procedure. Data from both CPS and catheterization measurements will be analyzed to assess agreement. No investigational treatment or additional follow-up visits are required.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled for clinically indicated right heart catheterization
* Ability to provide informed consent

Exclusion Criteria:

* Heart transplant recipients
* Patients with a left ventricular assist device (LVAD)
* Presence of external devices (e.g., Holter monitors) or surgical scars/wounds that interfere with CPS measurements
* Measurement concerns related to data reliability or quality

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years and older who are scheduled to undergo clinically indicated right heart catheterization as part of their standard medical care. Participants will represent a diverse range of individuals with conditions requiring invasive hemodynamic assessment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac Performance System electronic data for Pulmonary Pressure | Single measurement prior to right heart catheterization
  Cardiac function metric measurement including Pulmonary Pressure measured in mmHg
Pulmonary artery catheter electronic data for Pulmonary Pressure | During right heart catheterization procedure
  Cardiac function metric measurement including Pulmonary Pressure measured in mmHg

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Huntsville Hospital Heart Center, Huntsville, Alabama
  - Endeavor Health, Evanston, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York
  - The Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Stern Cardiovascular Foundation, Inc. / Baptist Memorial Hospital, Germantown, Tennessee
  - Baylor College of Medicine, Houston, Texas